CLINICAL TRIAL: NCT05640115
Title: DECOMPRESS (DECompressing Obstruction of Malignancy: Percutaneous Renal vs Endoscopic Stent)
Brief Title: Obstruction of Malignancy: Percutaneous Renal vs Endoscopic Stent
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study stopped due to lack of accrual
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB22-0835
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Urinary Obstruction; Malignancy; Urinary Dysfunction; Ureter Obstruction; Ureter Injury
Keywords: urinary issues; urinary obstruction; cancer
MeSH Terms: conditions — Neoplasms; Ureteral Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Ureteral Stenting) (Experimental): Group A: Participants in this group will receive a standard of care ureteral stenting performed by a urologist.
  Interventions: Device: Ureteral Stent
- Group B (Percutaneous Nephrostomy) (Experimental): Participants in this group will receive a standard of care percutaneous nephrostomy tube placement performed by an interventional radiologist.
  Interventions: Device: Percutaneous Nephrostomy Tube Placement

INTERVENTIONS:
Device: Ureteral Stent — A ureteral stent is a soft, hollow tube that is placed temporarily into the ureter. The stent allows the urine to drain. The stent has a coil on each end that keeps it from moving. The top end coils in the kidney and the lower end coils inside the bladder.
  Arms: Group A (Ureteral Stenting)
Device: Percutaneous Nephrostomy Tube Placement — A percutaneous nephrostomy is the placement of a small, flexible rubber tube (catheter) through your skin into your kidney to drain your urine. It is inserted through your back or flank.
  Arms: Group B (Percutaneous Nephrostomy)

SUMMARY:
This research study will compare two procedures commonly used to treat urinary obstruction due to cancer. Sometimes cancer blocks one or both ureters (narrow tubes in the body that carry urine from the kidneys to the bladder). When these ureters become blocked, the body can no longer properly drain urine. This blocking of the ureters is called urinary obstruction, which can lead to kidney problems, infection, and pain. Treatment options for urinary obstruction include ureteral stent placement and percutaneous nephrostomy tube placement. Both treatment options require a doctor to place soft tubes (like a catheter) inside the body to help the ureters properly drain urine. These two treatment options have different success rates, risks, and effects on quality of life. By doing this study, researchers hope to learn which treatment option is best for individuals who develop urinary obstruction because of cancer. Participation in this research will last about 3 months.

DETAILED DESCRIPTION:
This research study will compare two procedures commonly used to treat urinary obstruction due to cancer. Sometimes cancer blocks one or both ureters (narrow tubes in the body that carry urine from the kidneys to the bladder). When these ureters become blocked, the body can no longer properly drain urine. This blocking of the ureters is called urinary obstruction, which can lead to kidney problems, infection, and pain.

Treatment options for urinary obstruction include ureteral stent placement and percutaneous nephrostomy tube placement. Both treatment options require a doctor to place soft tubes inside the body to help the ureters properly drain urine. A ureteral stent is an internal drainage tube allowing urine to drain from your kidney down to your bladder. The percutaneous nephrostomy tube is a tube that comes out your back that drains urine into a bag. These two treatment options have different success rates, risks, and effects on quality of life. By doing this study, researchers hope to learn which treatment option is best for individuals who develop urinary obstruction due to cancer. Participation in this research will last about 3 months.

If you agree to participate:

* The study doctor will not pick which one of the two treatments described above you will receive. We will use a computer to place you in one of the two study groups. The group the computer picks is by chance, like a flip of a coin. This is also called "randomization." You will have an equal chance of being in either group.
* You will receive either a retrograde ureteral stent or a percutaneous nephrostomy tube. A member of the research team will tell you which of the two treatments you will get, after the selection has been made.

ELIGIBILITY:
Inclusion Criteria

* Patients must have unilateral or bilateral hydronephrosis secondary to extrinsic compression by malignancy on cross sectional imaging.
* Age ≥18 years.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Anticoagulation that cannot be safely reversed in the peri-procedural time period.
* History of severe allergy to contrast media.
* Prior stent or nephrostomy in previous 6 months.
* Urethral or ureteric stricture disease.
* Lower urinary tract structural abnormalities or urinary diversion precluding retrograde ureteral stent placement.
* On blood pressure support or clinically unstable.
* Pregnant women are excluded from this study because the radiation from either procedure is known to have the potential for teratogenic or abortifacient effects.
* Previous renal transplant.
* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Trial Feasibility (as assessed by number of enrolled and recruited patients) | 3 months
  The feasibility of a definitive randomized trial, specifically to quantify patient willingness to be randomly assigned treatment with retrograde ureteral stent versus percutaneous nephrostomy tube placement for malignant ureteral obstruction. The number of patient eligible and subsequent recruitment rates. Feasibility will be defined as successfully enrolling 50 patients in the 12 month enrollment period.

SECONDARY OUTCOMES:
Rate of Success for Participants Randomized to Percutaneous Nephrostomy vs. Ureteral Stent Placement | 6 months
  The rate of technical success when randomizing patients to percutaneous nephrostomy or ureteral stent placement for managing malignant ureteral obstruction. This rate of technical success will be assessed by:
  * Decompression failure (defined as any of the following: technical failure of study procedure, stable or worsening hydronephrosis on imaging at 3 months follow up, urosepsis within 3 months of procedure, or need for additional decompression procedure (stent or nephrostomy placement) within 2 months after initial procedure
  * Adverse surgical events (defined as grade ≥3 Clavien-Dindo classification)
  * Patient reported outcomes at baseline, 7-day, 30-day and 90-day post-procedure using the Brief Pain Inventory, PROMIS Adult Physical Function Short Form (v2.0), and American Urological Association Symptom Score
  * Compliance rate with questionnaires
  * Reasons for non-randomisation, percentage of non-consenting participants who choose nephrostomy vs. retrograde ureteral stenting

CONTACTS AND LOCATIONS:
Overall Officials: Parth Modi, MD, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF